CLINICAL TRIAL: NCT02175459
Title: Investigating Predictive Factors of Diabetes Occurence After Duodenalpancreatectomy
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Joslin Diabetes Center (Other); University of Siena (Other); University of Copenhagen (Other); Istituto di Neuroscienze Consiglio Nazionale delle Ricerche (Network); University of Pisa (Other)
Responsible Party: Principal Investigator, Giaccari Andrea, associate professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 14081985
Record Dates: First submitted 2014-06-23; First posted 2014-06-26 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: GLUCOSE METABOLISM; DIABETES; PANCREATIC ISLETS; Exocrine Pancreatic Dysfunction; Exocrine Pancreas Conditions; Exocrine Pancreatic Insufficiency; Endocrine Pancreas Disorder
Keywords: Beta cell function; Islet cell crosstalk; Incretin intraislet System; Biomarkers; MiRNA; ncRNA; Pancreatic exocrine endocrine crosstalk; Diabetes of exocrine pancreas
MeSH Terms: conditions — Diabetes Mellitus; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — PANCREAS SAMPLES
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Regeneration of mature cells that produce functional insulin represents a major focus of current diabetes research aimed at restoring beta cell mass in patients with most forms of diabetes. The capacity to adapt in response to diverse physiological conditions during life and the consequent ability to cope for increased metabolic demands is a distinctive feature of the endocrine pancreas in the regulation of glucose homeostasis. Both beta and alpha cells are dynamically regulated to continually maintain a balance between proliferation, neogenesis, and apoptosis. In this proposal, the investigators will focus on exploring key mechanism(s) that potentially regulate islet cell plasticity in altered glucose metabolic states.

Investigators will explore in a unique cohort of individuals who undergo duodenal pancretectomy. Prior to their surgery will be performed in vivo studies (Hyperglycemic clamp, Euglycemic Hyperinsulinemic clamp and Mixed Meal Tests) to accurately assess glucose homeostasis parameters to classify each individual into metabolic phenotypes. Then exploit the opportunity to collect pancreas samples from these patients who will be evaluated again after surgery, the investigators will determine the ability of the remnant pancreas to compensate for the acute reduction in islet mass and perform correlations between ex vivo and in vivo parameters.

Specifically, the patients will be subjected to incretin secretion (mixed meal), metabolic status (OGTT), insulin secretion characteristics (first and second phase responses), β-cell insulin content evaluation (arginine bolus). Subsequently, pancreas samples will be evaluated for morphometry, and proteomics and gene expression analyses of islet cell samples obtain by laser capture will allow a detailed investigation of mechanisms that contribute to islet plasticity. The overall goal of this project is to investigate key mechanisms driving the ability of islet mass to adapt to diverse metabolic states. We aim to explore modifications in gene expression and proteomics and correlate them with specific metabolic phenotypes, in order to determine key regulators of islet morphology.

ELIGIBILITY:
Inclusion Criteria:

* SCHEDULED FOR PANCREATECTOMY
* NO DIABETIC and DIABETIC

Exclusion Criteria:

* CHRONIC DESEASES
* STEROID THERAPY

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective pancreaticoduodenectomy for periampullary neoplasms will be enrolled in the study. Indications for surgery will be periampullary neoplasms, i.e.
  tumors of the Vater's ampulla, distal CBD and periampullary duodenum. Patients with pancreatic cancer will be excluded from the study. The metabolic features of all patients will be assessed before and after surgery. The patients will visit the Division of Endocrinology for studies at least 1 week before surgery. Only patients with normal cardiopulmonary and kidney functions, as determined by medical history, physical examination, screening blood tests, electrocardiogram and urinalysis, and not on any antidiabetic medications will be enrolled for metabolic assessments before and after surgery. Each subject will undergo, on separate days, a hyperinsulinemic euglycemic clamp, a hyperglycemic clamp and a mixed meal test one week before and after a variable period of recovery from the surgical procedure.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in metabolic status (normal glucose tolerance, impaired glucose tolerance, diabetes) | baseline, 1 month after surgery and 1year after surgery
  Metabolic status will be determined with oral glucose tolerance test and patients will be classified according their metabolic status (after 1 month and 1 year after surgery).

SECONDARY OUTCOMES:
Changes in incretin levels from baseline | baseline, 1 months after surgery and 1 year after surgery
  Incretin levels (GLP1 and GIP) will be measured during mixed meal test.
Change in insulin secretion from baseline | baseline, 1 month after surgery and 1 year after surgery
  Insulin secretion will be measured by Hyperglicemic clamp.
islet cell areas (beta, Alpha and delta cell positive area) | baseline
  Pancreas section will be immunostained for insulin, glucagon and somatostatin and Each section will be analyzed separately by measuring total insulin, glucagon or somatostatin positive areas, as well as the total pancreas section area, using Image Pro Plus software version 4. 5.1 . The β, α or δ cell areas will be expressed as percentage of total pancreas section area.
changes in beta cell function in the context of disease of exocrine pancreas | baseline
  Insulin secretion will be measured by Hyperglicemic clamp and ogtt.
changes in intraislet ncRNA in different metabolic status | baseline
  ncRNA sequenting in plasma and pancreas samples

OTHER OUTCOMES:
change in gene expression analysis among different groups of baseline metabolic status | baseline
  Extract of islet cells will be dissected from pancreatic sections by laser capture microdissection and then extracted RNA will be analyzed by real time PCR analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology - Catholic University, Rome, RM, Italy

REFERENCES:
- [Derived] Quero G, Laterza V, Di Giuseppe G, Lucinato C, Massimiani G, Nista EC, Sionne F, Biffoni B, Brunetti M, Rosa F, De Sio D, Ciccarelli G, Fiorillo C, Menghi R, Langellotti L, Soldovieri L, Gasbarrini A, Pontecorvi A, Giaccari A, Alfieri S, Tondolo V, Mezza T. A single-center prospective analysis of the impact of glucose metabolism on pancreatic fistula onset after pancreaticoduodenectomy for periampullary tumors. Am J Surg. 2024 Dec;238:115987. doi: 10.1016/j.amjsurg.2024.115987. Epub 2024 Sep 24. PMID 39342881
- [Derived] Mezza T, Ferraro PM, Di Giuseppe G, Moffa S, Cefalo CM, Cinti F, Impronta F, Capece U, Quero G, Pontecorvi A, Mari A, Alfieri S, Giaccari A. Pancreaticoduodenectomy model demonstrates a fundamental role of dysfunctional beta cells in predicting diabetes. J Clin Invest. 2021 Jun 15;131(12):e146788. doi: 10.1172/JCI146788. PMID 33905373
- [Derived] Mezza T, Ferraro PM, Sun VA, Moffa S, Cefalo CMA, Quero G, Cinti F, Sorice GP, Pontecorvi A, Folli F, Mari A, Alfieri S, Giaccari A. Increased beta-Cell Workload Modulates Proinsulin-to-Insulin Ratio in Humans. Diabetes. 2018 Nov;67(11):2389-2396. doi: 10.2337/db18-0279. Epub 2018 Aug 21. PMID 30131390